CLINICAL TRIAL: NCT00167154
Title: Efficacy of Risperidone in the Management of Suicidality in Major Depressive Disorder
Brief Title: Risperidone and Suicidality in Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Roberta May, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F030929002; RIS-DED-402
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Depression
Keywords: suicidality; antipsychotic; antidepressant; treatment
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- risperidone (Experimental): risperidone
  Interventions: Drug: Risperidone and placebo comparator
- placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: Risperidone and placebo comparator

INTERVENTIONS:
Drug: Risperidone and placebo comparator — Up to 2 mg risperidone or matching placebo daily

SUMMARY:
The purpose of this trial is to investigate the efficacy of risperidone as an adjunct to an antidepressant treatment in the acute management of suicidality during an episode of major depressive disorder.

DETAILED DESCRIPTION:
Using a double blind, placebo-controlled design, subjects diagnosed with a current episode of major depressive disorder (defined by DSM-IV criteria and supported by the Mini International Neuropsychiatric Interview), severe with suicidality despite currently taking an antidepressant, will be enrolled in the eight-week study. The treatment will be initiated by randomizing patients to receive risperidone or placebo in addition to the antidepressant that the patient is already taking. The clinical efficacy will be evaluated after 4 days, weekly for 4 weeks, then every other week for 4 weeks with the efficacy measures. During the eight-week study, treatment with risperidone or placebo will continue at the highest effective dosage (up to 2 mg per day). The dose of the antidepressant will not be changed during the study.

ELIGIBILITY:
Inclusion Criteria:

1. 19-60 years of age
2. Diagnosis of major depressive disorder, currently severe with suicidality
3. A total score of Montgomery-Asberg Depression Rating Scale (MADRS) =/> 25 with the suicide sub-score =/> 4
4. Currently is taking an antidepressant at a therapeutic dose for longer than 3 weeks
5. In good physical health

Exclusion Criteria:

1. Depression without suicidality
2. Presence of major psychiatric conditions other than major depressive disorder, such as bipolar disorder, schizophrenia, or anxiety disorders (except for generalized anxiety disorder)
3. Depressive symptoms induced by alcohol or substance abuse
4. Psychotic features which are predominant at the initial evaluation
5. Unstable major medical illness, such as cardiac disease or diabetes
6. Female subjects who are pregnant, breastfeeding, or, if of child-bearing potential, unwilling to use adequate birth control measures

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2007-04 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
CGI | 8 weeks
  Clinical Global Impression

SECONDARY OUTCOMES:
MADRS | 8 weeks
  Montgomery Asberg Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Li, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Reeves H, Batra S, May RS, Zhang R, Dahl DC, Li X. Efficacy of risperidone augmentation to antidepressants in the management of suicidality in major depressive disorder: a randomized, double-blind, placebo-controlled pilot study. J Clin Psychiatry. 2008 Aug;69(8):1228-1236. doi: 10.4088/jcp.v69n0805. PMID 18681749